CLINICAL TRIAL: NCT00610688
Title: High Prevalence of Rickets and Subclinical Maternal and Childhood Vitamin D Deficiency in the Middle East: a Randomized Controlled Trial of Prenatal Vitamin D Supplementation to Prevent Vitamin D Deficiency in Mothers and Their Infants
Brief Title: Controlled Trial of Prenatal Vitamin D3 Supplementation to Prevent Vitamin D Deficiency in Mothers and Their Infants
Acronym: PA 03-103
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: United Arab Emirates University (Other); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2008-0931
Record Dates: First submitted 2007-12-27; First posted 2008-02-08 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Prenatal Care; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prenatal Vitamin D3 (Placebo Comparator): Arm will receive prenatal vitamin with 400IU of cholecalciferol (Vitamin D3)along with a placebo tablet containing 0IU of Vitamin D
  Interventions: Drug: Prenatal Vitamin
- 2 (Experimental): Arm will receive prenatal vitamin with 400IU of cholecalciferol (Vitamin D3)along with a tablet containing 1600IU of Cholecalciferol (Vitamin D3)
  Interventions: Drug: Prenatal Vitamin; Drug: Cholecalciferol (Vitamin D3)
- 3 (Experimental): Arm will receive prenatal vitamin with 400IU of cholecalciferol (Vitamin D3) along with a tablet containing 3600IU of Cholecalciferol (Vitamin D3).
  Interventions: Drug: Prenatal Vitamin; Drug: Cholecalciferol (Vitamin D3)

INTERVENTIONS:
Drug: Prenatal Vitamin — Once daily, prenatal vitamin containing 400IU of Vitamin D, until delivery
Drug: Cholecalciferol (Vitamin D3) — Once daily, 1600IU dose of Vitamin D from 12 weeks gestation to delivery
  Arms: 2
Drug: Cholecalciferol (Vitamin D3) — Once daily, 3600IU dose of Vitamin D, from 12 weeks until delivery
  Arms: 3

SUMMARY:
The purpose of this research study is to compare the effects of higher dose vitamin D with commonly recommended dose in pregnant women to see which is better in achieving and/or maintaining sufficient vitamin D blood levels during pregnancy and in newborn infants as well as improving growth in the infant.

DETAILED DESCRIPTION:
Three dosages of Vitamin D will be administered; 400IU, 2000IU and 4000IU per day to pregnant women starting at less than 16 week gestation continued until delivery. The dose will be provided using a randomized control method. Serum levels of 25 hydroxy D will be measured in mothers at 12, 16, 28 and delivery. Cord blood 25 hydroxy D and the infants' birthweight, length and head circumference will be measured at birth.

ELIGIBILITY:
Inclusion Criteria:

* Women who are within the ages of 18-45 years
* In good general health
* 12 weeks pregnant (based on last menstrual period)

Exclusion Criteria:

* Mothers with preexisting type I or type II diabetes
* Mothers with preexisting hypertension
* Mothers with preexisting parathyroid disease or uncontrolled thyroid disease
* Mothers with multiple fetuses (e.g., twins, triplets, etc.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adekunle Dawodu, MBBS, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Hussein F Saadi, MD, Principal Investigator — United Arab Emirates University
Locations (2):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States
- United Arab Emirated Unitersity, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

REFERENCES:
- [Background] Dawodu A, Agarwal M, Sankarankutty M, Hardy D, Kochiyil J, Badrinath P. Higher prevalence of vitamin D deficiency in mothers of rachitic than nonrachitic children. J Pediatr. 2005 Jul;147(1):109-11. doi: 10.1016/j.jpeds.2005.03.001. PMID 16027707
- [Background] Dawodu A, Agarwal M, Hossain M, Kochiyil J, Zayed R. Hypovitaminosis D and vitamin D deficiency in exclusively breast-feeding infants and their mothers in summer: a justification for vitamin D supplementation of breast-feeding infants. J Pediatr. 2003 Feb;142(2):169-73. doi: 10.1067/mpd.2003.63. PMID 12584539
- [Background] Saadi HF, Dawodu A, Afandi BO, Zayed R, Benedict S, Nagelkerke N. Efficacy of daily and monthly high-dose calciferol in vitamin D-deficient nulliparous and lactating women. Am J Clin Nutr. 2007 Jun;85(6):1565-71. doi: 10.1093/ajcn/85.6.1565. PMID 17556694
- [Background] Dawodu A, Wagner CL. Mother-child vitamin D deficiency: an international perspective. Arch Dis Child. 2007 Sep;92(9):737-40. doi: 10.1136/adc.2007.122689. PMID 17715433
- [Background] Wagner CL, Taylor SN, Dawodu A, Johnson DD, Hollis BW. Vitamin D and its role during pregnancy in attaining optimal health of mother and fetus. Nutrients. 2012 Mar;4(3):208-30. doi: 10.3390/nu4030208. Epub 2012 Mar 21. PMID 22666547
- [Background] Dawodu A, Tsang RC. Maternal vitamin D status: effect on milk vitamin D content and vitamin D status of breastfeeding infants. Adv Nutr. 2012 May 1;3(3):353-61. doi: 10.3945/an.111.000950. PMID 22585912
- [Background] Dawodu A, Wagner CL. Prevention of vitamin D deficiency in mothers and infants worldwide - a paradigm shift. Paediatr Int Child Health. 2012 Feb;32(1):3-13. doi: 10.1179/1465328111Y.0000000024. PMID 22525442
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Dawodu A, Saadi HF, Bekdache G, Javed Y, Altaye M, Hollis BW. Randomized controlled trial (RCT) of vitamin D supplementation in pregnancy in a population with endemic vitamin D deficiency. J Clin Endocrinol Metab. 2013 Jun;98(6):2337-46. doi: 10.1210/jc.2013-1154. Epub 2013 Apr 4. PMID 23559082

RESULTS

PARTICIPANT FLOW:
Groups:
- 400 IU: Arm will receive prenatal vitamin with 400IU of Vitamin D along with a placebo tablet containing 0IU of Vitamin D
- 2000 IU: Arm will receive prenatal vitamin with 400IU of Vitamin D along with a tablet containing 1600IU of Vitamin D
- 4000 IU: Arm will receive prenatal vitamin with 400IU of Vitamin D along with a tablet containing 3600IU of Vitamin D
Period: Overall Study
Arm/Group | 400 IU | 2000 IU | 4000 IU
Started | 64 | 65 | 63
Completed | 55 | 52 | 55
Not Completed | 9 | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 IU | 2000 IU | 4000 IU | Total
Number analyzed (Participants) | 64 | 65 | 63 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 64 | 65 | 63 | 192
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (5.5) | 27.4 (4.8) | 25.7 (5.5) | 26.9 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 63 | 192
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Arab Emirates | 64 | 65 | 63 | 192
Maternal serum 25 hydroxy Vitamin D (25(OH)D) [Mean (Standard Deviation); unit: nmol/L] | 21.5 (13.0) | 20.5 (11.9) | 19.6 (7.7) | 20.7 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Maternal Serum and Neonatal Serum 25-hydroxyvitamin D Measurement
Description: Maternal serum 25-hydroxyvitamin D measurement at 12, 16, 28 weeks during pregnancy and at delivery and cord blood or neonatal serum 25-hydroxyvitamin D measurement
Time Frame: 12, 16, 28 weeks and at maternal delivery and neonatal birth
Population: Intention to treat analysis.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | 400 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 55 | 52 | 55
nmol/L
  Maternal at 12 Weeks | 21.5 (1.6) | 20.5 (1.5) | 19.6 (1.0)
  Maternal at 16 Weeks | 40.7 (2.1) | 53.7 (2.3) | 60.7 (3.3)
  Maternal at 28 Weeks | 53.9 (3.2) | 82.3 (4.4) | 88.2 (4.2)
  Maternal at Delivery | 48.2 (3.1) | 64.9 (4.0) | 89.8 (4.6)
  Neonatal at Birth | 36.9 (2.8) | 48.3 (3.5) | 66.1 (3.2)

2. Secondary Outcome: Growth of the Newborn Infant as Measured by Crown-heel Length and Head Circumference at Birth
Description: Growth of the newborn infant as measured by crown-heel length in centimeters and head circumference in centimeters at birth
Time Frame: At delivery
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 400 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 55 | 52 | 55
cm
  Heel Crown Length | 51.9 (2.2) | 51.6 (2.8) | 50.9 (3.7)
  Head Circumference | 34.1 (1.4) | 34.5 (2.0) | 33.9 (2.2)

3. Secondary Outcome: Birthweight of Newborn Infant
Description: Growth of the Newborn Infant as Measured by Birthweight in grams.
Time Frame: Measured at birth.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | 400 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 55 | 52 | 55
Grams | 3100 (374) | 3191 (492) | 3103 (639)

ADVERSE EVENTS:
Arm/Group | 400 IU | 2000 IU | 4000 IU
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/65 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/65 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes